CLINICAL TRIAL: NCT04136496
Title: Evaluation of a Novel Axillary Lymph Node Ink Localization Technique: A Feasibility Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never activated / began due to hospital staff and resources being re-allocated to support the demands of the Covid-19 global pandemic.
Sponsor: The Ottawa Hospital (Other)
Responsible Party: Principal Investigator, Dr. Raman Verma, Principal Investigator, The Ottawa Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180569-01H
Record Dates: First submitted 2019-10-02; First posted 2019-10-23 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer; Axillary Lymphadenitis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Study A: 10-20 patients Study B: 25-50 patients
  Study B will incorporate more patients as this is the population which we are more interested in, and will benefit the greatest from this technique. Study A is to determine if it is technically feasible and obtain feedback from the surgeons
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ink placed before chemotherapy (Study A) (Active Comparator): In Study A, 0.5 mL of Black Eye Ink will be placed in the metastatic LN after neoadjuvant therapy
  Interventions: Device: Black-Eye Ink
- Ink placed after chemotherapy (Study B) (Active Comparator): In Study B, 0.5 mL of Black Eye Ink will be placed before neoadjuvant therapy
  Interventions: Device: Black-Eye Ink

INTERVENTIONS:
Device: Black-Eye Ink — There are two proposed studies utilizing the Ink during differing timepoints.Both will identify patients with breast cancer, with a biopsied metastatic axillary lymph node(LN) with a tissue marker clip placed, as is current practice. In Study A, 0.5mL of Black Eye Ink will be placed in the metastatic LN after neoadjuvant therapy. In Study B, 0.5mL of Black Eye Ink will be placed before neoadjuvant therapy. In both studies, the LN containing the tissue marker clip will be the one to have the radioactive seed and Ink inserted. The seed will still be inserted, in the event the dye is not well-visualized. In both studies, the surgeon will attempt to find the LN by direct visualization and then confirm the appropriate LN has been removed by using the Gamma probe and intra-operative radiographs. If the seed is not within the tattooed node, the LN containing the seed will also be removed. All lymph nodes injected with Ink will be removed by the surgeon;no Ink-injected node remains in body.

SUMMARY:
Patients with breast cancer and metastatic axillary lymphadenopathy routinely undergo neo-adjuvant chemotherapy. For these patients, biopsy clip markers are inserted into the biopsy proven metastatic lymph node pre-treatment, as they may reach complete clinical response post-therapy. Limited axillary surgery, as opposed to a full axillary dissection, may then be indicated. It is still necessary to surgically excise the biopsy proven metastatic lymph node to accurately assess the pathologic response to therapy, and subsequently tailor post-surgical therapies appropriately. As such, these lymph nodes require pre-operative localization which, at The Ottawa Hospital, currently requires radioactive seed insertion under sonographic guidance, typically performed within 5 days of surgery. The procedure is often challenging, as both normal appearing lymph nodes and 3 mm biopsy clip markers are difficult and in some cases impossible, to visualize on ultrasound. At the time of surgery, the excised lymph node is radiographed, to ensure the radioactive seed and biopsy clip marker are both successfully excised. Localization with Ink has the potential to replace both the biopsy clip markers and radioactive seeds as the surgeons are able to directly visualize the Ink intra-operatively and excise the Inked lymph node. A preliminary study out of Stanford on 28 patients who underwent localization of axillary lymph nodes with Ink injected 1-211 days pre-operatively, in the pre neo-adjuvant and post neo-adjuvant settings, showed that lymph nodes injected with Ink are visible intra-operatively months after surgery, suggesting that this is a feasible localization technique (1).

ELIGIBILITY:
Inclusion Criteria:

* English or French speaking female patients, with a personal history of current pathologically proven breast cancer, over the age of 18 years [patients <18 would be considered a rare occurrence]
* Patients who will be undergoing neoadjuvant chemotherapy
* Patients who will be undergoing axillary lymph node radioactive seed localization
* Patients who will be undergoing axillary surgery

Exclusion Criteria:

* Allergic reaction to Black Eye Ink or any of its components
* Pregnancy
* Confirmed metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Identification rate of Inked nodes, containing seed and clip | 3 years
Identification rate of Inked nodes, not containing seed | 3 years
Identification rate of Inked nodes, not containing clip | 3 years
Identification rate of Inked nodes, not containing seed or clip | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Only study staff will have access to the study data. Only de-identified data will be collected in all study documents. The OHSN-REB and OHRI may review original patient medical records and relevant study records under the supervision of the investigator for audit purposes.